CLINICAL TRIAL: NCT06036953
Title: Effect of 8-week Frequency-specific Electrical Muscle Stimulation Combined With Resistance Exercise Training on Muscle Mass, Strength, and Body Composition in Men and Women: A Feasibility and Safety Study
Brief Title: Electrical Muscle Stimulation on Muscle Mass, Strength, and Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chi-Chang Huang, Distinguished Professor, National Taiwan Sport University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21-034-A2
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Electrical Muscle Stimulation; Exercise; Resistance Training
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No EMS (No Intervention)
- EMS (Experimental)
  Interventions: Device: electrical muscle stimulation

INTERVENTIONS:
Device: electrical muscle stimulation — The electric muscle stimulator (EMS) used in this study was from Funcare (Funcare Co., Ltd, Taichung, Taiwan). EMS electrodes were attached to the biceps of both hands, the abdomen, and the quadriceps of both legs sequentially. Each part was stimulated once a day for 30 minutes.
  Arms: EMS

SUMMARY:
In recent years, electrical muscle stimulation (EMS) devices have been developed as a complementary training technique that is novel, attractive, and time-saving for physical fitness and rehabilitation. While it is known that EMS training can improve muscle mass and strength, most studies have focused on the elderly or specific patient populations. The aim of this study was to investigate the effects of frequency-specific EMS combined with resistance exercise training for 8 weeks on muscle mass, strength, power, body composition, and parameters related to exercise fatigue. Additionally, we aimed to evaluate the feasibility and safety of EMS as an exercise aid to improve body composition. We recruited 14 male and 14 female subjects who were randomly assigned to two groups with gender parity (7 male and 7 female/group): (1) no EMS group and (2) daily EMS group. Blood biochemical routine analysis was performed every 4 weeks from pre-intervention to post-intervention, and body composition, muscle strength, and explosive power were evaluated 8 weeks before and after the intervention. We also performed an exercise challenge analysis of fatigue biochemical indicators after 8 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* smoking or drinking habits
* cardiovascular disease
* neuromuscular disease
* metabolic disease
* asthma
* pregnancy
* body mass index (BMI) over 27

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
VO2max | After 8 weeks of EMS
  To evaluate the maximum oxygen consumption and exercise performance, we used a treadmill (Pulsar, h/p/cosmos, Nussdorf-Traunstein, Germany) and an automatic breathing analyzer (Vmax 29c, Sensor Medics, Yorba Linda, CA, USA). In addition, a polar heart rate device was used to monitor the heart rate (HR). The speed range of the treadmill was set to 7.2 km/h and increased by 1.8 km/h every 2 min until fatigue, according to Bruce's protocol. When the breathing exchange rate (the volume ratio of carbon dioxide produced to oxygen consumed, VCO2/VO2) was higher than 1.10 and reached the maximum heart rate (maximum heart rate = 220 - age), oxygen consumption was considered to be maximum. The three highest VO2max peak were averaged to obtain the VO2max values of the individual volunteers.
Body composition_body fat | up to 8 weeks
  The multi-frequency principle was applied to measure body composition by using a bioelectrical impedance analyzer (BIA) on an InBody 570 device (In-body, Seoul, South Korea). To perform the measurements, after the subjects' palms and soles were removed from the sensors, the subjects stood on the footing electrodes and held the sensing handles with two hands. During the measurements, the subjects kept their arms open and left their bodies at an angle of 30° without speaking or moving. The subjects also fasted for at least 8 h before the test. The body fat were meansure
Body composition_muscle mass | up to 8 weeks
  The multi-frequency principle was applied to measure body composition by using a bioelectrical impedance analyzer (BIA) on an InBody 570 device (In-body, Seoul, South Korea). To perform the measurements, after the subjects' palms and soles were removed from the sensors, the subjects stood on the footing electrodes and held the sensing handles with two hands. During the measurements, the subjects kept their arms open and left their bodies at an angle of 30° without speaking or moving. The subjects also fasted for at least 8 h before the test. The muscle mass were meansure
Grip strength | up to 8 weeks
  Use the armed grip machine (T.K.K.5401, Takei Scientific Instruments Co.,Ltd, Niigata, Japan) to measure, hold each of the left and right hands three times until they are weak, and record the maximum value
The Countermovement Jump (CMJ) Test | up to 8 weeks
  The CMJ test is a practical, effective, reliable, and simple method of measuring lower limb strength, which is related to the maximum speed, strength and explosive force of the lower limbs. For this test, participants stood on the Kistler force measurement platform (9260AA, Kistler Co., Ltd., Switzerland) on both feet and performed to inspection. During the test, they were asked to put their hands on their hips and remain on the platform. After that, they were asked to squat down until the knees bent 90 degrees and then to immediately jump as high as possible. The average power (MF), were recorded during the jump. Each participant repeated the test 3 times, and CMJ data were obtained at the designated points. The instrument was calibrated for each individual's weight.
Clinical Biochemistry of lactate level | After 8 weeks of EMS
  For assessment of fatigue-related indices, volunteers fasted for at least 8 h before the 60% VO2max fixed intensity exercise challenge. Blood samples were collected with an arm venous catheter at indicated time points during exercise and recovery periods, including baseline (0), 30 (E30) min during the exercise phase, and 60 (R60) min in the recovery phase. Serum lactate (mmol/L), were assessed for monitoring physiological adaptation. All biochemical indices were assessed using an autoanalyzer (Hitachi 7060, Tokyo, Japan).
Clinical Biochemistry of ammonia level | After 8 weeks of EMS
  For assessment of fatigue-related indices, volunteers fasted for at least 8 h before the 60% VO2max fixed intensity exercise challenge. Blood samples were collected with an arm venous catheter at indicated time points during exercise and recovery periods, including baseline (0), 30 (E30) min during the exercise phase, and 60 (R60) min in the recovery phase. Serum ammonia (umol/L), were assessed for monitoring physiological adaptation. All biochemical indices were assessed using an autoanalyzer (Hitachi 7060, Tokyo, Japan).
Clinical Biochemistry of glucose level | After 8 weeks of EMS
  For assessment of fatigue-related indices, volunteers fasted for at least 8 h before the 60% VO2max fixed intensity exercise challenge. Blood samples were collected with an arm venous catheter at indicated time points during exercise and recovery periods, including baseline (0), 30 (E30) min during the exercise phase, and 60 (R60) min in the recovery phase. Serum glucose (mg/dL), were assessed for monitoring physiological adaptation. All biochemical indices were assessed using an autoanalyzer (Hitachi 7060, Tokyo, Japan).

SECONDARY OUTCOMES:
Safety assessment - AST | baseline, 4 week and 8 week
  Safety is assessed function of liver such as AST (8-38 IU/L).
Safety assessment - ALT | baseline, 4 week and 8 week
  Safety is assessed function of liver such as ALT (4-44 IU/L).
Safety assessment - BUN | baseline, 4 week and 8 week
  Safety is assessed function of kidney such as Bun (6-20 mg/dl)
Safety assessment - Creatinine | baseline, 4 week and 8 week
  Safety is assessed function of kidney such as Creatinine (0.6-1.3 mg/dl)
Safety assessment - Uric Acid | baseline, 4 week and 8 week
  Safety is assessed function of kidney such as Uric Acid (3.4-7.6 mg/dl)
Safety assessment - total protein | baseline, 4 week and 8 week
  Safety is assessed function of kidney such as total protein (6.4-8.9 g/dl)
Safety assessment - free fatty acid | baseline, 4 week and 8 week
  Safety is assessed function of lipid metabolism such as free fatty acid (0.1-0.9 mmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Graduate Institute of Sports Science, National Taiwan Sport University, Taoyuan District, Taiwan